CLINICAL TRIAL: NCT06797778
Title: Oral Health Promotion Program in Schools in Polígono Sur
Acronym: OHPPSPS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Antonia Domínguez Reyes, Full Professor Faculty of Dentistry, University of Seville
Other Study IDs: 0059-N23
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Educational and Preventive Session for Dental Caries; Oral Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this observational study is to evaluate oral health before and after conducting an educational session on oral hygiene in schoolchildren from 3 schools in the Polígono Sur of Seville.

The main questions it aims to answer are:

* To find out the needs of schoolchildren for oral treatment.
* To analyse whether the educational sessions carried out serve to improve the oral health of schoolchildren.

The researchers will compare the results of different academic years to see if it serves to improve.

The participants are examined at the school during the school year. The educational sessions are carried out at the school during the school year.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren whose legal guardians agree to participate

Exclusion Criteria:

* Schoolchildren whose legal guardians do not consent to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Preschool and primary school children in schools in Polígono Sur.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental caries | pre-intervention and immediately after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Sevilla, Seville, Sevilla, Spain